CLINICAL TRIAL: NCT02896634
Title: Use of Dried Blood Spot for Clinical Mass Spectrometry Analysis
Brief Title: Analysis by Clinical Mass Spectrometry of Bloodstains
Acronym: BUVAMASS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: SPOT-TO-LAB Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: 9622
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Patient Blood Biobank

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Dried whole blood spots on filter paper and plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- group with inflammation: Selection of samples from biobank with groups with inflammation
  Interventions: Biological: clinical biology analyzes spectrometry mass
- group with denutrition: Selection of samples from biobank with groups with denutrition
  Interventions: Biological: clinical biology analyzes spectrometry mass
- group with none: Selection of samples from biobank with groups with none
  Interventions: Biological: clinical biology analyzes spectrometry mass
- group with both: Selection of samples from biobank with groups with both.
  Interventions: Biological: clinical biology analyzes spectrometry mass

INTERVENTIONS:
Biological: clinical biology analyzes spectrometry mass — clinical biology analyzes spectrometry mass

SUMMARY:
Dried Blood Spot or DBS is a collection of blood capillary drops spotted and dried on to a filter paper used for different bioanalysis. In comparison to conventional blood testing, DBS offers practical, analytical, clinical and financial advantages. This less invasive sampling is already used in infectious diseases screening and is useful for persons with poor venous (babies, drug users or elderly). Mass-spectrometry-based analyses allow protein quantification on very low amount of blood sample. In the project we combine the two approaches to measure on DBS blood proteins with clinical relevance -including many FDA approves biomarkers). The detection of the relevant clinical analytes will be validated on available patient samples in accordance with the clinical norm ISO15189 and the requirement for CE IVD marking. This will allow commercial developments (kits, protocols...) realized with the industrial partner Spot-to-lab

DETAILED DESCRIPTION:
Analyses of blood spotted and dried on a matrix (DBS), has been used since the 1960s in clinical chemistry neonatal screening. Since then, many clinical analytes, including nucleic acids, small molecules and lipids, have been successfully measured using DBS.

DBS collection is in fact less invasive than classical venous puncture, it can be carried out by the patient at home and shipped by regular mail with no particular risk of contamination. The use of DBS in routine for the detection of transmissible diseases, as well as for the follow-up of chronic disease like diabetes, represent a safer and less costly evolution of clinical biology for the society.

However the routine use of DBS is yet is limited. The major limitations of using DBS are represented by the small blood volumes associated with DBS sampling (5-10 μL) and by the limited possibility to detect peptides and proteins.

In this program, we will address this issue by adapting to DBS mass spectrometry (MS) quantification of proteins/peptides. This relies on the detection of distinctive proteotypic peptides (peptides which sequence is specific to a unique protein). The specificity of such assays using triple quadrupole mass spectrometer is based on the capability to detect peptides by three molecular characteristics: retention time, precursor ion mass (m/z) and fragment ion mass (m/z). The combination of the precursor ion mass and the fragment ion mass z, highly specific, is called a transition. This approach is named when several peptides are detected in a single run "multiple reaction monitoring" or MRM. Using this approach, the direct analysis of the trypsin digest of blood samples is possible without additional sample fractionation.

In a series of preliminary experiments, we could detect on single DBS puch of 6mm of diameter, 35 plasma proteins. Several proteins are of clinical relevance such as apolipoprotein A, B, C, ceruloplasmin, haptoglobin, plasminogen, transthyretin (prealbumin) or serum albumin. We will extend the range of blood protein detected by MS. Focus will be put on select biomarkers to generate clinically relevant panels that can be used for patients monitoring, nutrition monitoring and for the follow-up of frailty in elderly people .

Innovative workflows to obtain more rapid, efficient and costless detection will be developed. We will also evaluate a new type of DBS card (Noviplex™) which collects plasma instead of whole blood, and is expected to achieve better clinical concordance of the results between DBS and classical sampling. The detection of the relevant clinical analytes will be validated on available patient samples in accordance with the clinical norm ISO15189 and the requirement for CE IVD marking. This will allow commercial developments (kits, protocols...) realized with the industrial partner Spot-to-lab. This start-up has already put on the market DBS analyses resulting from previous collaborative research. Being able to measure peptide/proteins from DBS in parallel with other clinical analytes also developed by Spot-To-Lab (vitamin D, HbA1c…) represents a breakthrough which will gives major perspective to the use of DBS in clinical chemistry for disease detection and monitoring.

ELIGIBILITY:
Inclusion criteria:

* Signature of informed consent to have their sample stored in a biobank and use for research.
* Having a standard blood test scheduled during their consultation or hospitalization.

Exclusion criteria:

- Lack of informed and signed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be selected in a biobank from patients in neurology and geriatry units who gave their informed consent. Samples will be represented by leftover from blood sampling realized for the care and the determination of the concentration of blood analytes, including, albumin and CRP.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
clinical biology analyzes spectrometry mass | 1 day
  clinical biology analyzes spectrometry mass

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Lehmann, PH PU, Study Director — UHMONTPLLIER
Locations (1):
- LEHMANN, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided